CLINICAL TRIAL: NCT01980329
Title: Polymorphic Effects of Cytochrome P450 3A5 on Pharmacokinetics of Maraviroc and Its Metabolites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Namandjé N. Bumpus, PhD, Assistant Professor, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NA_00078492
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Cytochrome P450 CYP3A5 Enzyme Polymorphism; Healthy Subjects; Pharmacokinetics of Maraviroc
Keywords: CYP3A5; maraviroc; polymorphism
MeSH Terms: interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Maraviroc (Experimental): single oral administration of 300 mg maraviroc
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc
  Other Names: Selzentry

SUMMARY:
The purpose of this study is to evaluate the influence of genetic polymorphism of cytochrome P450 3A5 on pharmacokinetics of maraviroc and its oxidative metabolites

DETAILED DESCRIPTION:
This study aims to evaluate the effects of CYP3A5 genotype on pharmacokinetics of maraviroc and its oxidative metabolites. A single oral dose of 300 mg maraviroc will be given to 24 eligible healthy individuals who will be screened and determined to have specific CYP3A5 genotype - 8 homozygous wild type (2 CYP3A5*1 alleles), 8 heterozygous (1 CYP3A5*1 allele and 1 mutant allele), and 8 without wild type genotype (2 mutant alleles). Blood samples will be drawn and urine samples will be collected immediately before and during a 32-hr period following the dose. The concentrations of maraviroc and its oxidative metabolites from the blood and urine samples will be measured and the pharmacokinetics of maraviroc and its metabolites will be compared among the three groups with different CYP3A5 polymorphic status.

--------------------------------------------------------------------------------

ELIGIBILITY:
Inclusion Criteria:

* Healthy with no acute medical illness
* Willing to provide written informed consent
* Age 18-65 years
* Negative serum pregnancy test (females only) at screening and a negative urine pregnancy test (females only) on day of dosing
* HIV seronegative at screening, as determined by any licensed ELISA
* At screening, no evidence of hepatic or renal impairment (LFT's < 1.5 Upper Limit of Normal (ULN), creatinine clearance > than 60 ml/min, total bilirubin below ULN, AST and ALT below 1.5 ULN)
* 8 subjects with homozygous CYP3A5 allele *1 (wild type)
* 8 subjects with 1 CYP3A5*1 allele and 1 mutant allele
* 8 subjects with CYP3A5 allele other than *1

Exclusion Criteria:

* Concomitant medication (prescription or over-the-counter) or herbal supplements for which there is a known risk of pharmacokinetic or pharmacodynamic drug interactions, including those that inhibit CYP3A4 as listed on the P450 Drug Interaction Table (http://medicine.iupui.edu/clinpharm/ddis/table.aspx)
* History of postural hypotension or cardiovascular disease
* Active medical or psychological condition that, in the opinion of the investigator, might put the volunteer at undue risk or interfere with the participation of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve | 0-32 hour post dose administration

SECONDARY OUTCOMES:
Clearance | 0-32 hr post dose administration
Plasma peak concentration | 0-32 hr post dose administration
Plasma half-life | 0-32 hr post dose administration
Urinary metabolic ratio | 0-32 hr post dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Namandje N Bumpus, Ph.D, Principal Investigator — Johns Hopkins University; Craig W Hendrix, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins University School of Medicine Division of Clinical Pharmacology, Baltimore, Maryland, United States